CLINICAL TRIAL: NCT03956004
Title: A Technology-enabled Decision Aid for Patients With Hip and Knee Osteoarthritis
Brief Title: The Impact of a Technology-enabled Decision Aid, for Patients With Hip and Knee Osteoarthritis on Decision Quality, Level of Shared Decision-making, Patient Satisfaction and Magnitude of Limitations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Kevin Bozic, Professor of Surgery, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018-11-0042
Record Dates: First submitted 2019-03-25; First posted 2019-05-20 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Osteoarthritis, Knee
Keywords: shared decision making; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Full decision aid, consisting of education on osteoarthritis and treatment options, preferences and values elicitation, and personalized risk/benefit estimates based on patient's response to patient-reported outcome measures.
  Interventions: Other: OM1 Dell Shared Decision Making Tool
- Control (Active Comparator): Education component of the decision aid only.
  Interventions: Other: Education material from OM1 Dell Shared Decision Making Tool

INTERVENTIONS:
Other: OM1 Dell Shared Decision Making Tool — Decision aid meant to improve shared decision making among patients and providers.
  Arms: Experimental
Other: Education material from OM1 Dell Shared Decision Making Tool — Investigator-written educational material and quiz to test knowledge of osteoarthritis and treatment options.
  Arms: Control

SUMMARY:
This study evaluates a technology-enabled decision aid that provides evidence-based education (i.e. on understanding the condition, treatment options and comparisons, patient values and question & answer quiz) and personalized, quantifiable benefit-risk ratio alongside the level of potential benefit in relation to joint stiffness, joint pain and quality of life. The study will be performed in the setting of an integrated care system providing patient-centered care for hip and knee osteoarthritis over the full cycle of care. The impact of a technology-enabled decision aid incorporating predictive analytics with machine learning capabilities on decision quality, activation, experience & limitations of patients in this setting is relatively unknown.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a presumptive diagnosis of knee OA aged between 45 and 89 (in-line with the decision aid algorithm)
* Radiographic evidence of moderate to severe osteoarthritis (Kellgren and Lawrence grade 3-4)
* KOOS Jr scores between 0-85 (in-line with the decision-aid algorithm)
* Participant able to give informed consent for participation in the study

Exclusion Criteria:

* Kellgren and Lawrence scale for classification of osteoarthritis grade 0-2
* Patients with a prior experience of total joint replacement
* Patient with experience with the pilot form of the decision aid
* Patients undergoing consideration for revision joint replacement
* Patients seeking care for trauma condition or psoriatic/rheumatoid arthritis
* Non-English or Non-Spanish speakers
* Patients with BMI below 20 or above 46 (in-line with the decision-aid algorithm)

Ages: 45 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Knee Osteoarthritis Decision Quality Instrument | Day 1
  Decision process subscore. Participants receive 1 point for a response of "yes" or "a lot/some." The total points are summed and then divided by the total number of items to result in scores from 0-100%, with higher scores indicated a more shared decision making process.
Knee Osteoarthritis Decision Quality Instrument | Day 1
  Concordance subscore (A summary score (0-100%) indicating the percentage of patients who received treatment that matched their stated preference will be generated.)

SECONDARY OUTCOMES:
CollaboRATE | Day 1
  Level of shared decision making. Range of 0-9. Higher scores represent more shared decision making.
Numeric rating scale-satisfaction | Day 1
  Patient satisfaction with management of condition. Range of 0-10 with 0 representing complete dissatisfaction and 10 representing complete satisfaction.
Knee injury and osteoarthritis outcome score, joint replacement (KOOS JR) | 6 months after baseline visit
  Measure of patient-reported, knee-related stiffness, pain, and function. Raw score range 0-28, converted to interval score of 0-100, where 0 represents total knee disability and 100 represents perfect knee health.
Undergoing joint replacement surgery or not | Day 1
  Decision to undergo total knee replacement surgery (yes/no). Obtained by asking provider or through medical record note.
Average time of patient visit and average time spent with provider | Day 1
  Minutes. Time of entire visit will be recorded in addition to time spent with primary provider.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Bozic, Principal Investigator — University of Texas at Austin
Locations (1):
- UT Health Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jayakumar P, Moore MG, Furlough KA, Uhler LM, Andrawis JP, Koenig KM, Aksan N, Rathouz PJ, Bozic KJ. Comparison of an Artificial Intelligence-Enabled Patient Decision Aid vs Educational Material on Decision Quality, Shared Decision-Making, Patient Experience, and Functional Outcomes in Adults With Knee Osteoarthritis: A Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e2037107. doi: 10.1001/jamanetworkopen.2020.37107. PMID 33599773